CLINICAL TRIAL: NCT01871974
Title: Phase I Study of FK949E - Multiple Dose Study of Non-Elderly Adult Patients With Major Depressive Disorder (MDD)
Brief Title: Study to Evaluate Safety and Tolerability of FK949E in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6949-CL-0001
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder Patients
Keywords: FK949E; Antipsychotic; Quetiapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-dose group FK949E (Experimental): oral
  Interventions: Drug: FK949E
- high-dose group FK949E (Experimental): oral
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — oral
  Other Names: extended release formulation of quetiapine

SUMMARY:
The objective of the study was to evaluate the safety and plasma concentration changes of quetiapine after multiple oral administration of FK949E (extended-release formulation of quetiapine) in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is a dose-titration study. In low-dose-group, patients receive prescribed dose on Day 5 after 3-step dose increases. In high-dose-group patients receive prescribed dose on Day 7 after 4-step dose increases. Patients receive prescribed dose of FK949E for 7 days in each group. The dosage period is 12 days in low dose group and 14 days in high dose group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder according to the DSM-IV-TR (Text Revision of the Diagnostic and Statistical Manual of Mental Disorders version-4)
* Female patients of childbearing potential with a negative serum pregnancy test result and who were willing and able to use a reliable method of birth control during the study
* Patients who could understand and comply with the requirements of the study, as judged by the investigator/sub-investigator

Exclusion Criteria:

* A current or past history of a DSM-IV-TR Axis I disorder other than major depressive disorder within 6 months prior to the study
* Diagnosis of a DSM-IV-TR Axis II disorder that was considered to have a major impact on the patient's current psychiatric status
* A history of substance or alcohol abuse or dependence excluding caffeine and nicotine
* Patients who were unable to abstain from drugs that induce or inhibit the drug-metabolizing enzyme CYP3A4 from 14 days prior to the start of study drug administration and throughout the study period
* Pregnant or lactating women
* Patients showing evidence or signs of renal or hepatic failure, serious heart disease, cerebrovascular disease, viral hepatitis B or C, or acquired immunodeficiency syndrome (AIDS) (carrier)
* A clinical finding that in the opinion of the investigator/sub-investigator could be negatively affected by the study or that would affect the study results (e.g., hypertension, unstable angina)
* Conditions that could affect absorption and metabolism of the study medication (e.g., malabsorption syndrome, liver disease)
* A current diagnosis of malignant tumor unless in remission for at least 5 years (except basal or squamous cell skin carcinoma)
* A current or past diagnosis of transient ischemic attack (TIA)
* A history of seizure disorder, except for febrile convulsions
* Application of electroconvulsive therapy within 90 days prior to the start of study drug administration
* Use of a depot antipsychotic injection and inability to be off the drug for a period of twice the dosing interval prior to the start of study drug administration and throughout the study period
* Patients could require psychotherapy (other than supportive psychotherapy) during the study period, unless psychotherapy had been ongoing for a minimum of 90 days prior to the start of study drug administration
* A score of ≥ 3 on the HAM-D17 Item (suicide) or a suicide attempt within the past 6 months, and those judged to be at serious suicidal or homicidal risk in the opinion of the investigator/sub-investigator
* A current or past history of diabetes mellitus* or glycated hemoglobin (HbA1c) of ≥ 6.5% at screening within 2 months before the start of study drug administration (*refer to the guidelines for monitoring blood glucose levels in patients treated with atypical antipsychotics)
* A white blood cell count (WBC) of ≤ 3,000/mm3 at screening assessment
* Elevation of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values at screening assessment (grade 2 or higher according to the "Criteria for Classification of the Grade of Adverse Drug Reactions to Pharmaceutical Products" (Pharmaceutical Affairs Bureau Safety Division's Notification No. 80 issued on 29 June 1992))
* A known history of hypersensitivity to quetiapine or to any other component in the FK949E tablets at the time of providing written informed consent
* Treatment with quetiapine for depressive symptoms or bipolar disorder (mania) at the time of providing written informed consent
* Participation in another clinical study or post-marketing study within 12 weeks prior to the start of study drug administration

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of unchanged quetiapine | For 24 hours after dosing

SECONDARY OUTCOMES:
AUC (area under the curve) of unchanged quetiapine | For 24 hours after dosing
tmax of plasma concentration of unchanged quetiapine | For 24 hours after dosing
t1/2 of plasma concentration of unchanged quetiapine | For 24 hours after dosing
Safety assessed by the incidence of adverse events, clinical lab tests, vital signs, 12-lead ECGs and physical exam | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kansai
  - Kantou

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=177